CLINICAL TRIAL: NCT01981421
Title: Usefulness of Multi-parametric, Quantitative MR Imaging for Staging of Hepatic Fibrosis in the Patients With Chronic Hepatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0193
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Liver Fibrosis
Keywords: Liver fibrosis; Elastography; MR Elastography; Quantitative imaging
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver fibrosis: patients who had chronic liver disease

SUMMARY:
Liver fibrosis has been considered as irreversible change. However, recent study showed that early stage liver fibrosis could be reversible and a lot of new drugs are now developing or developed including anti-viral treatment. Liver biopsy is considered as golden standard for the evaluation of liver fibrosis. But biopsy specimen through biopsy only consists of 1/50000 of the whole liver and heterogeneity of liver fibrosis, accurate diagnosis of liver fibrosis is still challenging. Furthermore, its invasive nature, repeated biopsy is practically almost impossible. Hence, non-invasive diagnosis of liver fibrosis is important. In this study we hypothesized that multi-parametric MR imaging including MR elastography, conventional DWI, and IVIM can predict changes of liver stiffness after anti-viral therapy in patients with chronic liver disease. We will enroll 60 biopsy-proven patients and perform multi-parametric MR imaging at the enrollment and one year later to evaluate changes in quantitative values in MR.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had chronic hepatitis
* Patients who underwent liver biopsy within 6 months
* Patients older than 18 years old

Exclusion Criteria:

* patient who had pregnancy
* patient 18 or below 18 years old

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have chronic liver disease and who are planned to receive anti-viral treatment.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes in quantitative values measured from Multi-parametric MRI before and after anti-viral treatment | 1 year after enrollment
  Elasticity, conventional ADC value, IVIM ADC value, T2* value, T1 rho value will be compared before and after anti-viral treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Yonsei University Health System, Seoul, South Korea